CLINICAL TRIAL: NCT01547403
Title: Evaluation of Customer Support Issues, Questions, or Alleged Complaints Regarding Use of Approved Commercially Distributed Scout DS Product in the Field
Brief Title: Customer Support Response Study
Acronym: CUSTOM
Status: Withdrawn | Type: Observational
Why Stopped: Protocol no longer meeting sponsor objectives
Sponsor: VeraLight, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: VL-2719
Record Dates: First submitted 2012-02-27; First posted 2012-03-07 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes
Keywords: Screening for Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary objective of the CUSTOM study is to respond to customer support issues (outside of the US) and to assess the impact of a particular treatment or perturbation relative to an initial control measurement. Sequential subject measurements will be analyzed to determine if a given action or condition induces a score shift, an inflation of measurement variance or elevated outlier rates.

DETAILED DESCRIPTION:
The SCOUT DS device is not yet approved by the FDA for sale in the United States, but currently is being marketed in Canada and other countries. Customers who are using the device have contacted the sponsor with questions about testing conditions which might affect the reproducibility of measurements.

The objective is to obtain information to allow the Sponsor to address these issues. The concerns fall into three broad categories:

• Factors affecting the interface between the skin and the test sensor

These would include the effects of skin care products applied to the forearm, subject activity that changes perfusion to the skin and subject movement during the test procedure.

* General operating conditions Issues such as ambient temperature, lighting, and height of the table on which the SCOUT DS device rests have been questioned as possible factors influencing accuracy.
* Rare subject disorders

Included here would be subject skin abnormalities or physiologic changes which occur so infrequently that they were not well represented in previous data sets. Examples of such rare conditions would include scleroderma, capillary angiomata, and Raynaud phenomenon.

ELIGIBILITY:
Inclusion Criteria:

* Males and/or females greater than or equal to 18 years of age

Exclusion Criteria:

* Have received investigational treatments in the past 14 days
* Have psychosocial issues that interfere with an ability to follow study procedures
* Are known to be pregnant
* Have scars, tattoos, rashes or other disruption/discoloration on the left volar forearm.
* Have been treated on the past month with oral steroid therapy or topical steroids applied to the left forearm. Inhaled steroid therapy is not a basis for exclusion
* Are receiving medications that fluoresce (A list of excluded medications is located in Appendix H)
* Are known to have, or at risk for, photosensitivity reactions (e.g., sensitive to ultraviolet light, or taking medication known to cause photosensitivity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Up to 500 volunteers age 18 and above, of either sex and of any ethnic background, will be recruited at one site.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint for CUSTOM Trial | Up to 1 year
  The primary objective of the CUSTOM study is to respond to customer support issues and to assess the impact of a particular treatment or perturbation relative to an initial control measurement. Sequential subject measurements will be analyzed to determine if a given action or condition induces a score shift.
  Subjects will undergo measurements and a diabetes risk score is generated from the SCOUT device. The scale of the score is 0-100. Subjects are not provided with this score as the device is still investigational in the US.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Aase, MD, Principal Investigator — VeraLight, Inc.
Locations (1):
- VeraLight, Albuquerque, New Mexico, United States